CLINICAL TRIAL: NCT00000812
Title: A Phase I, Placebo-Controlled, Dose-Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Thalidomide in Subjects With HIV-1 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 267; 42,240; 11243 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Thalidomide
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
PRIMARY: To evaluate the safety, tolerability, and pharmacokinetics of daily oral thalidomide.

SECONDARY: To examine the effect of thalidomide on antiviral activity and tumor necrosis factor-alpha (TNF-alpha) production, and the correlation between TNF-alpha inhibition and viral burden.

A protein in the blood called tumor necrosis factor (TNF-alpha) is abnormally elevated in patients with HIV infection and may cause the body to produce more virus. In vitro studies have demonstrated that thalidomide reduces TNF-alpha levels and inhibits production of HIV. However, more information on the pharmacological and immunological aspects of thalidomide is needed.

DETAILED DESCRIPTION:
A protein in the blood called tumor necrosis factor (TNF-alpha) is abnormally elevated in patients with HIV infection and may cause the body to produce more virus. In vitro studies have demonstrated that thalidomide reduces TNF-alpha levels and inhibits production of HIV. However, more information on the pharmacological and immunological aspects of thalidomide is needed.

Patients are randomized to receive oral thalidomide or matching placebo (3:1) at one of three dose levels daily for 8 weeks. All 12 patients at a dose level must receive treatment for at least 2 weeks before dose escalation in subsequent patients occurs. The MTD is defined as the dose level immediately below that at which 3 or more of 9 patients receiving thalidomide experience dose-limiting toxicity. Patients are followed for a total of 16 weeks.

PER 6/20/95 AMENDMENT: Patients in cohort 1 should discontinue the previous 50 mg formulation of thalidomide once the new formulation is available. Those patients may either wash out for 4 weeks and recommence the study or discontinue the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed for occasional use (chronic use is permitted only if clinician deems that medication can be discontinued in the event of overlapping toxicity):

* CNS active agents, such as alcohol, narcotics (i.e., morphine, codeine, meperidine), barbiturates, benzodiazepines, tricyclic antidepressants, phenothiazines, sedating antihistamines, or over-the-counter sleeping aids.

Patients must have:

* HIV infection.
* CD4 count 200 - 500 cells/mm3.
* No active opportunistic infection requiring systemic therapy within the past 14 days.
* NOTE: Women must be post-menopausal or provide written documentation of surgical sterilization, and sexually active men must use a barrier method of contraception, beginning 4 weeks prior to study entry and continuing until 4 weeks following end of treatment.

PER AMENDMENT 8/2/96:

* Been on stable licensed antiretroviral treatment for 60 days prior to study entry or must not have received any antiretroviral medications for 60 days prior to study entry.

Prior Medication:

Required:

* Patients must have been on stable licensed antiretroviral treatment for 60 days prior to study entry or must not have received any antiretroviral medications for 60 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy requiring chemotherapy.
* Grade 2 or worse peripheral neuropathy.
* Medical condition that would interfere with evaluation of patient.

Concurrent Medication:

Excluded in all patients:

* Didanosine ( ddI ).
* Zalcitabine ( ddC ).
* Stavudine ( d4T ).
* Other immunologically active agents.
* Systemic cytotoxic chemotherapy.

Excluded in all patients unless taken only occasionally or unless medication could be stopped in the event of overlapping toxicity:

* CNS active agents, such as alcohol, narcotics (i.e., morphine, codeine, meperidine), barbiturates, benzodiazepines, tricyclic antidepressants, phenothiazines, sedating antihistamines, or over-the-counter sleeping aids.

Patients with the following prior conditions are excluded:

* History of active tuberculosis within 3 months prior to study entry.
* History of intolerance to thalidomide such as fever, rash, or neuropathy.

Prior Medication:

Excluded within 14 days prior to study entry:

* Systemic chemotherapy.

Excluded within 30 days prior to study entry:

* Topical, oral, and systemic corticosteroids.
* Pentoxifylline.
* Interferons.
* Interleukins.
* Cimetidines.
* Acetylcysteine or other glutathione depleting agents.
* Other putative immunomodulatory agents such as thymosin alpha 1, thymopentin, isoprinosine, ditiocarb sodium, ampligen, and immune globulin.

PER AMENDMENT 8/2/96:

Excluded within 60 days prior to study entry:

* Therapy with investigational antiretroviral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teppler H, Study Chair; Pomerantz R, Study Chair
Locations (6):
- United States (6):
  - University of Colorado Hospital CRS, Aurora, Colorado
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Wohl D, Pomerantz R, Schmitz J, Aweeka F, Fox L, Weng D, Spritzler J, Robinson W, Holohan M, Teppler H. Thalidomide pharmacokinetics (PK) safety and effect on HIV viral load and immune parameters. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 352)
- [Background] Wohl DA, Aweeka FT, Schmitz J, Pomerantz R, Cherng DW, Spritzler J, Fox L, Simpson D, Bell D, Holohan MK, Thomas S, Robinson W, Kaplan G, Teppler H; National Institute of Allergy and Infectious Diseases AIDS Clinical Trials Group 267. Safety, tolerability, and pharmacokinetic effects of thalidomide in patients infected with human immunodeficiency virus: AIDS Clinical Trials Group 267. J Infect Dis. 2002 May 1;185(9):1359-63. doi: 10.1086/340133. Epub 2002 Apr 16. PMID 12001058